CLINICAL TRIAL: NCT04667286
Title: Pronation in Spontaneously Breathing Patients With Acute Respiratory Failure Deu to Covid-19: Multicenter, Randomised Study
Brief Title: Awake Pronation for Covid-19 Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Azienda USL Reggio Emilia - IRCCS (Other Government); Azienda Ospedaliera di Bolzano (Other); Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, dr. Stefano Nava, professor and chief of respiratory and critical care unit, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1117/2020/Sper/AOUBo
Record Dates: First submitted 2020-12-11; First posted 2020-12-14 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Covid-19 Infection
MeSH Terms: conditions — COVID-19 | interventions — Prone Position

STUDY DESIGN:
Intervention Model Description: randomised trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygen and Prone Position (PP) (Experimental): Oxygen via a Venturi mask in order to keep an oxygen saturation between 92 and 96% plus PP for a minimum of 10 hrs a day
  Interventions: Procedure: Prone Position (PP)
- Oxygen (Active Comparator): Oxygen via a Venturi mask in order to keep an oxygen saturation between 92 and 96%
  Interventions: Procedure: Prone Position (PP)

INTERVENTIONS:
Procedure: Prone Position (PP) — Prone the patients on oxygen for at least 10 hrs a day

SUMMARY:
Observational studies have shown that prone position (PP) in spontaneously breathing patients, may improve oxygenation in individuals with Acute Respiratory Failure (ARF), due to Covid-19 infection.

None so far have evaluated the clinical efficacy of this approach on the patients' outcomes and in a randomised control fashion

DETAILED DESCRIPTION:
Observational studies have shown that prone position (PP) in spontaneously breathing patients, may improve oxygenation in individuals with Acute Respiratory Failure (ARF), due to Covid-19 infection.

These studies were mainly physiological and reported in a subset of patients a poor tolerance. Indeed most of the beneficial effects on gas exchage disappeared in around 40% of tyhe patients, once the patients regained the supine position.

None so far have evaluated the clinical efficacy of this approach on the patients' outcomes and in a randomised control fashion.

This holds particularly true in those patients affected by mild de-novo ARF (PaO2/FiO2 ratio within the range of 200-300), where any form of respiratory support like Continuous Positive Airways Pressure (CPAP), High Flow Nasal Cannula (HFNC) or Noninvasive ventilation (NIV), may be not yet indicated, especially if the patients are admitted to a regular ward as for the case of Covid-19 pandemics, due to the lack of "protected" beds.

ELIGIBILITY:
Inclusion Criteria:

* confirmed COVID-19 infection using PCR
* Acute Respiratory Failure ( 200 <PaO2/FiO2 <300) and respiratory rate < 30 atti/min
* O2 therapy initiated <72 hrs
* informed consent

Exclusion Criteria:

* Glasgow Coma Scale (GCS) < 13
* pH< 7,45, PaCO2 >45 mmHg
* need for HFNC, CPAP, NIV or intubation
* hemodynamic instability increase of 80-90 mmHg or reduction of 30-40 mmHg in systolic blood pressure
* severe arrythmia of myocardial infarction
* need for sedation
* intolerance to PP
* pregnancy
* Body mass index (BMI) > 35 kg/m2.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-16 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
number of day free of ventilatory support | 1 month
  number of days in which the patient will not need (according to standardized criterai) any for of these ventilatory support like NIV,CPAP, HFNC or intubation

SECONDARY OUTCOMES:
changes in respiratory pattern | 1 month
  recording of tidal volume (when possible) and respiratory frequency
daily changes in the ratio SaO2/FiO2 | 1 month
  Daily changes in oxygen saturation (SaO2) and Fraction of Inspired Oxygen (FiO2)
dyspnea | 1 month
  using a dedicated scale (i.e. Borg numbered from 0 to 10)
comfort during PP | 1 month
  using a dedicated visual analog scale (VAS with a lenght of 20 cm)

OTHER OUTCOMES:
number of hours on PP | 1 month
  recording of the actual time spent in PP

CONTACTS AND LOCATIONS:
Overall Officials: stefano nava, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (3):
- Italy (3):
  - Sant'Orsola Malpighi, Bologna
  - Bolzano Hospital, Bolzano
  - University of Modena, Modena

IPD SHARING:
Plan to Share IPD: No